CLINICAL TRIAL: NCT05171530
Title: An Exploratory Clinical Study of Lenvatinib Combined With Single-agent Taxanes as Second-line Therapy for the Treatment of HER2-negative Advanced Gastric Cancer
Brief Title: Lenvatinib With Taxane Drugs Treatment for Advanced Gastric Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Yan Shi, Associate Professor, Ruijin Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LOGIC
Record Dates: First submitted 2021-12-05; First posted 2021-12-29 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: HER2-negative Advanced Gastric Cancer
MeSH Terms: interventions — lenvatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lenvatinib with taxane drugs treatment for advanced gastric cancer (Experimental): Experimental: Lenvatinib plus taxane drugs The subjects in this arm will receive a Lenvatinib combined with single-agent taxanes therapy. A standard dose of chemotherapy: paclitaxel 135mg/m2 every 3 weeks or docetaxel 75mg/m2 every 3 weeks will be administrated. Lenvatinib is exploring four doses of 4mg, 8mg, 12mg, and 16mg, orally once a day every 3 weeks. In the first cycle, lenvatinib was administered 5 days before chemotherapy，once a day. Chemotherapy lasts up to 6 cycles, and lenvatinib continues to be administered until the disease progresses, intolerable side effects, or death.
  Subjects will be enrolled serially. For subject safety, the preceding subject must have completed therapy and there is no obvious DLT within 21 days before the next subject can be treated.
  Interventions:
  * Drug: Paclitaxel or Docetaxel
  * Drug: Lenvatinib
  Interventions: Drug: Lenvatinib plus taxane drugs

INTERVENTIONS:
Drug: Lenvatinib plus taxane drugs — * Drug: Paclitaxel Dose: 135mg/m2 Other Name: PTX
  * Drug: Docetaxel Dose: 75mg/m2 Other Name: FA
  * Drug: Lenvatinib Dose: 4mg, 8mg, 12mg,16mg Other Name: FA

SUMMARY:
The goal of this clinical trial is to study the safety and efficacy of lenvatinib combined with single-agent taxanes therapy in patients with HER2-negative advanced gastric cancer that have failed at the standard first-line therapy.

DETAILED DESCRIPTION:
This study is being conducted to establish safety and preliminary efficacy of Lenvatinib plus taxane drugs treatment for HER2-negative advanced gastric cancer after failure of first-line treatment.

The study will adopt the "3+3" dose escalation design. All patients received a standard dose of chemotherapy: paclitaxel 135mg/m2 every 3 weeks or docetaxel 75mg/m2 every 3 weeks. Lenvatinib is exploring four doses of 4mg, 8mg, 12mg, and 16mg, orally once a day every 3 weeks. In the first cycle, lenvatinib was administered 5 days before chemotherapy，once a day. Chemotherapy lasts up to 6 cycles, and lenvatinib continues to be administered until the disease progresses, intolerable side effects, or death.

In order to avoid the possible ineffectiveness caused by the patient being exposed to low doses, the initial dose of 4 mg was enrolled in 1 patient. If there is no obvious dose-limiting toxicity (DLT) after the first dose, the dose escalation adopts a "3+3" method from the 8mg dose: if none of the 3 subjects in the previous dose group has a DLT within 21 days, the next dose study will be carried out; if one subject in the group has DLT occurs, then 3 additional subjects should be added to the dose group; if the 3 subjects have 1 or more DLTs, the trial terminated and the previous dose was regarded as the maximum tolerated dose (MTD).

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and the willingness to provide written informed consent.
2. Advanced gastric cancer diagnosed by histopathological or cytological examination, no uncontrollable pleural and ascites;.
3. Age no less than 18 years.
4. Life expectancy greater than 3 months.
5. According to the RECIST (Response Evaluation Criteria in Solid Tumors) standard, there must be measurable lesions.
6. Failed at the standard first-line therapy, microsatellite stable (MSS) or no mismatch repair missing(PMMR), HER2 negative.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 .
8. Adequate liver/bone marrow function.
9. Female subjects must meet the following conditions: infertility or fertility and use high-efficiency contraceptive measures.
10. Male subjects agree to use approved contraceptive methods (e.g. birth control pills, barrier device, intrauterine device, abstinence) during the study and for 3 months following the last dose of the study cell infusion. Moreover, all men are absolutely prohibited from donating sperm within 1 year after receiving the last study treatment infusion.

Exclusion Criteria:

1. Previous use of lenvatinib or chemotherapy drugs in the regimen.
2. Pregnant or breast-feeding female, or not willing to take contraception measures during study.
3. Uncontrolled brain metastasis or mental illness.
4. Suffered from other uncured malignant tumors within the past 3 years or at the same time.
5. A history of active gastrointestinal bleeding within 3 months, incomplete obstruction or complete intestinal obstruction.
6. Uncontrollable high blood pressure are not suitable for enroll into the study.
7. Other uncontrolled diseases may cause abnormal death of the patient.
8. Untolerable liver/bone marrow function.
9. Factors that affect the administration of oral drugs (dysphagia, chronic diarrhea, complete intestinal obstruction, etc.
10. Previously allergic to the ingredients of the medicine in regimen.
11. Can't be followed up or obey protocol.
12. The investigator believes that it is not appropriate to participate in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2022-01-05 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 4 weeks after the last administration
  Incidence of DLT within 21 days of the first Lenvatinib application
Incidence of Treatment Related adverse events (TRAEs) | 4 weeks after the last administration
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
Incidence of dose-limiting toxicities (DLTs) | 4 weeks after the last administration
  All patients who have received at least one dose of treatment will be included in the safety analysis. Number of participants with dose-limiting toxicities as assessed by CTCAE v5.0
Incidence of Treatment Emergent Adverse Event (TEAEs) | 4 weeks after the last administration
  Number of participants with treatment emergent adverse events as assessed by CTCAE v5.0
Maximum tolerated dose of lenvatinib | 4 weeks after the last administration
  Maximum tolerated dose of lenvatinib in combination with single-agent chemotherapy

SECONDARY OUTCOMES:
Objective response rate (ORR) | up to 12 months
  Objective Response Rate is defined as the percentage of patients with a documented complete response or partial response (CR + PR) based on RECIST v1.1.
Disease control rate (DCR) based on the researcher's evaluation | up to 12 months
  Disease control Rate is defined as the percentage of patients with a documented complete response or partial response or stable disease (CR + PR+SD) based on RECIST v1.1.
Duration of Remission (DOR) based on the researcher's evaluation | up to 12 months
  The duration of remission (DOR) is defined as the time interval between the subject's first recording of disease remission to the first recording of disease progression.
Progression-free survival (PFS) based on the researcher's evaluation | up to 12 months
  Progression-free survival (PFS) is defined as the time interval from the first treatment of the subject to the first recording of disease progression or death due to any cause, whichever occurs first.
Overall survival (OS) | up to 12 months
  Overall survival is defined as the time from signing ICF until death from any cause.

OTHER OUTCOMES:
Exploratory Outcome | up to 8 weeks
  Dynamic contrast-enhanced ultrasound (DCE-US) was used to evaluate the the efficacy of anti-angiogenic therapy. Wash-in area under the curve (WiAUC) were quantitatively by DCE-US before the chemotherapy(d-4), d1 and 42 days after chemotherapy.
Exploratory Outcome | up to 8 weeks
  Mass spectrometry flow cytometry was used to detect the ratio and number of CD8+T cells on d0 and d42 after Lenvatinib therapy, and evaluates the correlation between changes in the immune microenvironment and the efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Shi, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No